CLINICAL TRIAL: NCT06323434
Title: Spinal CSF Leaks in Chronic Subdural Hematoma
Acronym: SPICE
Status: Recruiting | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Katharina Wolf, Clinician Scientist, University of Freiburg
Other Study IDs: spice1
Record Dates: First submitted 2024-01-05; First posted 2024-03-21 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Chronic Subdural Hematoma
Keywords: Spinal CSF leak; Spontaneous Intracranial Hypotension; CSF-venous fistula
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Cerebrospinal Fluid Otorrhea; Intracranial Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cSDH: 1. Chronic subdural hematoma on imaging (CT/MRI)
  2. Age: 18 years or older
  3. Informed consent

SUMMARY:
Background: Chronic subdural hematoma (cSDH) is a type of intracranial bleeding, predominantly affecting the elderly and males, with an estimated incidence of 8/100.000. The collection of subdural fluid expands slowly, leading eventually to brain tissue compression that results in neurological impairment such as seizures, cognitive decline, and paresis. Most patients need neurosurgical evacuation of the blood to improve and to prevent further, possibly permanent deterioration. Evidently, the cause of such a bleeding must be investigated and if possible treated, or preventive strategies need to be installed if possible. Spinal cerebrospinal fluid (CSF) leaks are a known cause of cSDH but are widely underdiagnosed in this population.

The spinal CSF leak causes CSF loss that leads to intracranial hypotension, expansion of intracerebral veins, and traction to the brain and the surrounding tissues. A cSDH is a severe complication of such a leak and occurs in about 30% of all cases with a predominance among the elderly. It is crucial to identify these patients with a spinal leak as treatment pathways differ essentially from patients without a leak. Some smaller studies indicated a prevalence of spinal CSF leaks among cSDH patients of 30% to 80% depending on selection criteria (age, extend of cSDH). Notably, the entity of the CSF-venous fistula, that has been discovered as recent as 9 years ago, and that by now is accounting for 20-25% of all spinal leaks, has not been considered in previous research on cSDH and spinal CSF leaks.

Currently, there is no prospective data on spinal CSF leaks in patients with cSDH. Establishment of such data is crucial to improve diagnostic and therapeutic algorithms for spinal CSF leaks in patients with cSDH.

Objective: To prospectively assess the prevalence of spinal CSF leaks in patients with cSDH Methods: This is a prospective observational, monocentric study on patients admitted due to cSDH to the Department of Neurosurgery at the Medical Center of the University of Freiburg. Treatment and diagnostic procedures will follow standard protocols. The number of spinal CSF leaks will be assessed to generate the prevalence of spinal CSF leaks in this patient cohort. Furthermore, clinical data, the specific type of the CSF leak, and imaging parameters are assessed systematically to estimate the diagnostic value of these measures.

DETAILED DESCRIPTION:
Background:

Chronic subdural hematoma (cSDH) refers to a blood- and fluid-collection between the brain and the dura that is most common in the elderly with a male predominance. Patients present with headaches, gait instabilities, cognitive impairments, decline of vigilance, hemiparesis, aphasia, or seizures. These symptoms usually lead to hospital admission where the diagnosis can be easily depicted by non-contrast computer tomography (CT), or magnetic resonance imaging (MRI). Image characteristics of the transformed hemoglobin of the blood indicate the chronicity, therefore, the rather slow development of this intracranial hemorrhage. Smaller parts of acute bleeding can attribute to a faster progression. Incidence across all ages is reported at about 8/100.000, while age-depended incidence increases up to 64/100.000 at age of > 79 years. About 2/3 present with unilateral, 1/3 with bilateral hematoma.

A symptomatic cSDH requires surgical treatment, which might range from twist drill trepanation with or without drain to open trepanation and fluid evacuation in order to prevent permanent brain damage and further deterioration. Recurrence rates are up to 20%. The mortality rate is increased even after successful treatment of the bleeding.

The actual cause for the development of cSDH is yet not sufficiently explored. While a history of minor head trauma is often reported as the leading cause of cSDH, a minor trauma cannot account for the entire pathology in cSDH. Some mechanisms are reported that are rather believed to maintain but not to initiate the process: Characteristic membranes are built that are thought to cause further exudation and hemorrhage. Fragile vessels are discussed to contribute to the process, stimulated by inflammation and poor angiogenesis. Recent efforts to therapeutically address inflammation as a primary target failed, which highlights the critical need of improved therapies.

Over the past years, it has become evident, yet widely neglected in clinical daily life, that many cases of cSDH are caused by spinal cerebro spinal fluid (CSF) leaks that lead to spontaneous intracranial hypotension (SIH). These leaks lead to a continuous loss of CSF, which therefore causes hypotension and traction within the skull that is most sever in upright position. This intracranial hypotension can lead to the development of cSDH.

If this underlying cause of cSDH is not diagnosed and if it remains untreated, the persistent spinal leak maintains the process of traction and bleeding - leading to a recurrence of the cSDH with a high likelihood and risking further brain damage. Also, there is a risk of further impairment of health and quality of life due to an untreated spinal CSF leak itself (e.g., chronic headache, hearing impairment up to hearing loss, cognitive decline, and superficial siderosis. Unfortunately, spinal CSF leaks are often not investigated, or overseen. The diagnostic sensitivity regarding spinal CSF leaks largely depends on the awareness, experience and dedication of the medical professionals. In an emergency due to intracranial bleeding, a medical history of seemingly fewer threatening symptoms like orthostatic headache or hearing impairment is likely overseen by patients and the medical team, alike. Thus, symptoms and signs are easily missed in cSDH cohorts if not specifically investigated.

In patients with atraumatic, bilateral cSDH, it has already become textbook knowledge that investigation for spinal CSF leaks should be conducted. Nevertheless, according to literature, current observations, and expert opinion, a limitation exclusively to bilateral cSDH cannot be justified and sets misdiagnosed patients at risk of further harm. It must be recognized that the mentioned limitation to bilateral cSDH is based on research at times of less sensitive diagnostics without knowledge on the variety of spinal CSF leaks. For example, the discovery of CSF-venous fistulas at the spine has been one of the few genuine new discoveries in Neuroradiology within the past 9 years. By now, within the investigator's cohort, this type of leak accounts for >20% of all leaks and is rather detected in the elderly (mean age 57 years vs. 44 years other leaks, p=0.002), a cohort that is also more likely to develop cSDH. For example: to investigate for CSF-venous fistulas, a conventional prone myelography would lead to a false-negative results, as myelography would need to be performed in lateral decubitus position. Furthermore, another type of a sacral leak has recently been discovered. Therefore, all formerly gathered data on cSDH and SIH need to be interpreted in respect to current developments and the former lack of diagnostic sensitivity. Thus, in experienced SIH centers, it has been established to screen for spinal leaks irrespective of age and size to prevent false treatment and recurrence of cSDH.

Literature on spinal CSF leaks in patients with bilateral and unilateral cSDH reports high rates ranging from 26% to even 80 %. The analysis of retrospective data of 216 SIH patients with a proven and surgically treated spinal CSF leak across all ages showed, that 60/216 (30%) had cSDH, with a clear predominance of bilateral (88%) over unilateral (12%) hematomas. Careful management of the bleeding and most importantly closure of the leak led - so far - to no detected recurrence of the cSDH in this cohort. Data also suggest that the development of cSDH is more likely in older SIH patients, which also are more likely to develop CSF-venous fistulas that yet have not been subject of investigation in cSDH cohorts. Also, the intake of oral anticoagulation should not prevent further investigation for spinal CSF leaks, as there is evidence that oral anticoagulation is quite often not the definitive cause of cSDH but rather an additional factor.

In summary, cSDH and SIH are interlinked. Older data suggested that only younger patients with cSDH and bilateral cSDH should be suspected to suffer from spinal leaks. In contrast, current data imply that spinal leaks can cause unilateral and bilateral cSDH at any age. On the other hand, there might be a publication bias as with any retrospective studies and prospective data is needed.

Aims:

Primary aim:

a) To estimate the prevalence of spinal CSF leaks in patients with chronic subdural hematoma (cSDH)

Secondary aims:

1. To estimate the proportion of different spinal CSF leak types in patients with chronic subdural hematoma (cSDH)
2. To investigate differences in the proportion of spinal CSF leaks and subtypes stratified by age, and stratified by sex
3. To investigate the proportion of interventions needed, delineate clinical parameters, diagnostic findings, resurge need, and differences in outcome in patients with and without proven spinal CSF leak in patients with chronic subdural hematoma (cSDH)
4. To evaluate the diagnostic value of clinical and diagnostic parameters to detect spinal CSF leak in patients with chronic subdural hematoma (cSDH)

Methods:

The study is monocentric. The design is prospective, longitudinal, and observational.

New patients with cSDH admitted to the investigator's department will be screened on a daily basis. The patients, or their caregivers, respectively, will be informed and included upon given written informed consent. As many patients will need emergency evacuation of the subdural hematoma, patients will be specifically asked to consent that data starting at time of admission can be investigated.

Diagnostic, treatment, and follow-up procedure will follow clinical standards according to established standard operating procedures (SOP). This standard includes a screening MRI of the brain and spine for signs of spinal CSF leaks. These results in combination with patients' history will be given to the interdisciplinary SIH-Board for consideration. In case of evidence for SIH, further investigation for spinal CSF leaks are initiated.

Evidence of SIH can be found in the MRI of the spine as spinal longitudinal epidural collection (SLEC) for some leak types. Further signs indicating a moderate or higher risk of a spinal CSF leaks is a Bern Score of 3 or higher in the MRI of the head. Also, clinical symptoms indicative of spinal CSF leaks, such as orthostatic headache are considered.

According to the SOP, the follow-up visits will be scheduled depending on the clinical course that determines the frequencies of visits needed. Follow-ups are conducted at least up to 6 months to scan for resurge of the cSDH and outcome of the procedures, including at least one follow-up visit including imaging after 3 months.

This study aims to collect a dataset containing clinical workups up to the 6 months follow-up per participant following standardoperating procedures.

Considerations on sample size As this is an explorative, observational study without formal sample size estimation, the study is limited by time of duration (24 months), not by exact numbers.

By an estimated population of 1.74 Mio and an incidence of cSDH of 8/100.000, about 140 patients should be expected per year, adding up to approximately 280 patients with cSDH. Considering some patients and/or caregivers who do not consent, a realistic number of 220 to 240 might be achieved.

With this sample size, it would be able to estimate the prevalence with a 95% Wilson confidence interval (CI) with a width of 11-13% (for prevalences of 20-80%). For example with a sample size of 220 and a prevalence of 50%, the 95% Wilson CI would be 43.4-56.5%.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic subdural hematoma on imaging (CT/MRI)
2. Age: 18 years or older
3. Informed consent

Exclusion Criteria:

1. General contraindications for MRI examination (e.g., pacemaker wearers, implanted insulin, or pain pump, neurostimulator, etc.)
2. Recurrent chronic subdural hematoma and previously performed diagnostics and treatment in compliance to the current cSDH SOP
3. Severe brain injury, acute subdural hematoma, epidural hematoma, subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Department of Neurosurgery with cSDH on imaging will be approached and informed about the study after initial treatment of the intracranial hemorrhage if indicated.
  In case of legal incapacity, the designated caregiver and legal council will be approached for consent. The inclusion of this vulnerable group is considerable as they represent an important subgroup of patients. Otherwise, the trial would not be suitable to represent a typical patient cohort, and data would not be meaningful for clinical standards. The inclusion of vulnerable groups seems justifiable as there will be no additional procedure performed other than clinical standard work-up.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
evidence of a spinal CSF leak (yes/no) | up to 4 weeks
  The primary endpoint is evidence of a spinal CSF leak (yes/no) in patients with chronic subdural hematoma (cSDH) depicted by MRI: evidence spinal longitudinal extradural fluid (SLEC), or Myelogram: detection of spinal CSF leak

SECONDARY OUTCOMES:
Number of identified CSF leak types: | up to 4 weeks
  * Ventral leak
  * Lateral leak
  * CSF-venous fistula
  * Sacral leak
  * Undefined
Number of diagnostic procedures performed: | up to 6 month
  * CT head
  * MRI head
  * MRI spine
  * Myelography
Number, and site of interventions needed for cSDH: | up to 6 month
  * Twist drill trephination
  * Twist drill trephination with drain
  * Conventional trepanation
  * Twist drill trephination or conventional trepanation with drain and any form of controlled lavage (saline and or clot lysis)
  * Embolisation of media meningeal artery
Color of hematoma evacuated: | up to 6 month
  * clear to amber-colored (yes/no)
  * "motor-oil" appearance (yes/no)
Age | at time of inclusion
  in years
body height | at time of inclusion
  height (m)
body weight | at time of inclusion
  weight (kg) Body mass index derived by height and weight (kg/m2)
Body mass index (BMI) | at time of inclusion
  derived by height and weight (kg/m2)
sex | at time of inclusion
  * male
  * female
  * diverse
Karnofsky Index | up to 6 months
  Range: 0-100%, 100% indicating best health
Anti-platelet therapy intake | up to 6 months
  * yes
  * no
Anticoagulation intake | up to 6 months
  * yes
  * no
Blood pressure medication intake | up to 6 months
  * yes
  * no
Lipid regulation medication intake | up to 6 months
  * yes
  * no
Hormonal regulation medication intake | up to 6 months
  * yes
  * no
Immunotherapeutic medication intake | up to 6 months
  * yes
  * no
other medication intake | up to 6 months
  * yes
  * no
history of trauma | up to 6 months
  * No trauma,
  * recent trauma within 0-4 weeks,
  * past trauma >4 weeks ago
national institutes of health stroke scale (NIHSS) | up to 6 months
  range 0 to 42, 0 indicating no neurological deficits
gait disorder | up to 6 months
  * yes
  * no
Modified Rankin Scale (mRS) | up to 6 months
  range 0-6, 0 indicating best health
Headache-Impact-Test (HIT)-6 | up to 6 months
  - Headache-Impact-Test (HIT)-6 range 36 to 78 points, 78 indicating highest impact of headaches
current working capacity, | up to 6 months
  range 0 to 5, 0 indicating full capacity
complaints | up to 6 months
  * current complaints (descriptively)
  * most stressful complaint (descriptively)
headache severity | up to 6 months
  range 0 to 10, 10 indicating most severe pain
Days within the last month | up to 6 months
  * with headaches
  * with pain medication intake in the last month
maximum duration being continuously upright | up to 6 months
  in hours
severeness of dizziness | up to 6 months
  - in 0 to 10, 10 being most severe
Severeness of shoulder- and neck pain | up to 6 months
  - in 0 to 10, 10 being most severe
severeness of nausea | up to 6 months
  - in 0 to 10, 10 being most severe
severeness of hearing disturbances and tinnitus | up to 6 months
  - in 0 to 10, 10 being most severe
severeness of cognitive deficits | up to 6 months
  - in 0 to 10, 10 being most severe
severeness of visual disturbances | up to 6 months
  - in 0 to 10, 10 being most severe
exhaustion | up to 6 months
  -rated between 0 to 5, with 5 indicating highest burden
ability to focus and concentrate | up to 6 months
  rated between 0 to 5, with 5 indicating highest burden
Patient's Global Impression of Change (PGIC) | up to 6 months
  Patient's Global Impression of Change (PGIC), range 7 to 42, 7 indicating highest improvements
Self-Administered Comorbidity Questionnaire (SCQ) | up to 6 months
  - 13-item Self-Administered Comorbidity Questionnaire (SCQ), range 0 to 39, 0 indicating lowest burden
5 dimension / 5 levels European Quality of life questionnaire (EQ-5D-5L) Index | up to 6 months
  <0 to 1, 1 indicating unimpaired health
5 dimension / 5 levels European Quality of life questionnaire (EQ-5D-5L) visual analogue scale | up to 6 months
  0 to 100, with 100 indicating unimpaired wellbeing
Hematocrit | up to 2 days
  in%
Size of the chronic subdural hematoma | up to 6 month
  mm^3
Volumetry of the cranial compartments | up to 6 month
  mm^3
Bern-Score according to Dobrocky et al | up to 6 month
  ange 0 to 9 with 9 indicating highest likelihood of a spinal CSF leak
  * Spinal longitudinal extradural fluid collection (SLEC)(yes/no)
  * DiverTICula (TIC) (yes/no)
Spinal longitudinal extradural fluid collection (SLEC) | up to 6 month
  * yes
  * no
DiverTICula (TIC) | up to 6 month
  * yes
  * no

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Beck, Prof., Principal Investigator — Department of Neurosurgery, Medical Center, University of Freiburg
Locations (1):
- University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck J, Gralla J, Fung C, Ulrich CT, Schucht P, Fichtner J, Andereggen L, Gosau M, Hattingen E, Gutbrod K, Z'Graggen WJ, Reinert M, Husler J, Ozdoba C, Raabe A. Spinal cerebrospinal fluid leak as the cause of chronic subdural hematomas in nongeriatric patients. J Neurosurg. 2014 Dec;121(6):1380-7. doi: 10.3171/2014.6.JNS14550. Epub 2014 Jul 18. PMID 25036203
- [Background] Dobrocky T, Grunder L, Breiding PS, Branca M, Limacher A, Mosimann PJ, Mordasini P, Zibold F, Haeni L, Jesse CM, Fung C, Raabe A, Ulrich CT, Gralla J, Beck J, Piechowiak EI. Assessing Spinal Cerebrospinal Fluid Leaks in Spontaneous Intracranial Hypotension With a Scoring System Based on Brain Magnetic Resonance Imaging Findings. JAMA Neurol. 2019 May 1;76(5):580-587. doi: 10.1001/jamaneurol.2018.4921. PMID 30776059
- [Background] Dumont TM, Rughani AI, Goeckes T, Tranmer BI. Chronic subdural hematoma: a sentinel health event. World Neurosurg. 2013 Dec;80(6):889-92. doi: 10.1016/j.wneu.2012.06.026. Epub 2012 Jun 19. PMID 22722034
- [Background] Edlmann E, Giorgi-Coll S, Whitfield PC, Carpenter KLH, Hutchinson PJ. Pathophysiology of chronic subdural haematoma: inflammation, angiogenesis and implications for pharmacotherapy. J Neuroinflammation. 2017 May 30;14(1):108. doi: 10.1186/s12974-017-0881-y. PMID 28558815
- [Background] El Rahal A, Beck J, Ahlborn P, Bernasconi C, Marbacher S, Wanderer S, Burkhardt JK, Daniel RT, Ferrari A, Hausmann O, Kamenova M, Kothbauer K, Lutz K, Mariani L, Alfieri A, Schoni D, Schucht P, Raabe A, Regli L, Kuhlen D, Seule M, Soleman J, Starnoni D, Zaldivar J, Zweifel C, Schaller K, Fung C. Incidence, therapy, and outcome in the management of chronic subdural hematoma in Switzerland: a population-based multicenter cohort study. Front Neurol. 2023 Sep 14;14:1206996. doi: 10.3389/fneur.2023.1206996. eCollection 2023. PMID 37780710
- [Background] Feghali J, Yang W, Huang J. Updates in Chronic Subdural Hematoma: Epidemiology, Etiology, Pathogenesis, Treatment, and Outcome. World Neurosurg. 2020 Sep;141:339-345. doi: 10.1016/j.wneu.2020.06.140. Epub 2020 Jun 25. PMID 32593768
- [Background] Hamou HA, Clusmann H, Schulz JB, Wiesmann M, Altiok E, Hollig A. Chronic Subdural Hematoma. Dtsch Arztebl Int. 2022 Mar 25;119(12):208-213. doi: 10.3238/arztebl.m2022.0144. PMID 35236548
- [Background] Hufschmidt, A., S. Rauer, F. Glocker, and Hrsg, eds. 2022. Neurologie compact. Stuttgart: Thieme und doi:10.1055/b000000096
- [Background] Kim HJ, Lee JW, Lee E, Kang Y, Ahn JM. Incidence of Spinal CSF Leakage on CT Myelography in Patients with Nontraumatic Intracranial Subdural Hematoma. Diagnostics (Basel). 2021 Dec 6;11(12):2278. doi: 10.3390/diagnostics11122278. PMID 34943515
- [Background] Kranz PG, Malinzak MD, Gray L, Willhite J, Amrhein TJ. Resisted Inspiration Improves Visualization of CSF-Venous Fistulas in Spontaneous Intracranial Hypotension. AJNR Am J Neuroradiol. 2023 Aug;44(8):994-998. doi: 10.3174/ajnr.A7927. Epub 2023 Jul 6. PMID 37414450
- [Background] Lutzen N, Aleman EB, El Rahal A, Volz F, Fung C, Beck J, Urbach H. Sacral Dural Tears as a Cause of Spontaneous Intracranial Hypotension. Clin Neuroradiol. 2023 Dec;33(4):957-964. doi: 10.1007/s00062-023-01292-0. Epub 2023 Jun 1. PMID 37261452
- [Background] Lutzen N, Beck J, Urbach H. Cerebrospinal Fluid Venous Fistula Imaging with Ultrahigh-Resolution Cone-Beam Computed Tomography. JAMA Neurol. 2023 Aug 1;80(8):870-871. doi: 10.1001/jamaneurol.2023.1640. PMID 37306975
- [Background] Mehta V, Harward SC, Sankey EW, Nayar G, Codd PJ. Evidence based diagnosis and management of chronic subdural hematoma: A review of the literature. J Clin Neurosci. 2018 Apr;50:7-15. doi: 10.1016/j.jocn.2018.01.050. Epub 2018 Feb 7. PMID 29428263
- [Background] Miah IP, Holl DC, Blaauw J, Lingsma HF, den Hertog HM, Jacobs B, Kruyt ND, van der Naalt J, Polinder S, Groen RJM, Kho KH, van Kooten F, Dirven CMF, Peul WC, Jellema K, Dammers R, van der Gaag NA; DECSA Collaborators. Dexamethasone versus Surgery for Chronic Subdural Hematoma. N Engl J Med. 2023 Jun 15;388(24):2230-2240. doi: 10.1056/NEJMoa2216767. PMID 37314705
- [Background] Miranda LB, Braxton E, Hobbs J, Quigley MR. Chronic subdural hematoma in the elderly: not a benign disease. J Neurosurg. 2011 Jan;114(1):72-6. doi: 10.3171/2010.8.JNS10298. Epub 2010 Sep 24. PMID 20868215
- [Background] Sahyouni R, Goshtasbi K, Mahmoodi A, Tran DK, Chen JW. Chronic Subdural Hematoma: A Historical and Clinical Perspective. World Neurosurg. 2017 Dec;108:948-953. doi: 10.1016/j.wneu.2017.09.064. Epub 2017 Sep 19. PMID 28935548
- [Background] Schievink WI, Maya MM, Barnard ZR, Moser FG, Jean-Pierre S, Waxman AD, Nuno M. Behavioral Variant Frontotemporal Dementia as a Serious Complication of Spontaneous Intracranial Hypotension. Oper Neurosurg. 2018 Nov 1;15(5):505-515. doi: 10.1093/ons/opy029. PMID 29534203
- [Background] Schievink WI, Maya MM, Harris J, Galvan J, Tache RB, Nuno M. Infratentorial Superficial Siderosis and Spontaneous Intracranial Hypotension. Ann Neurol. 2023 Jan;93(1):64-75. doi: 10.1002/ana.26521. Epub 2022 Oct 22. PMID 36200700
- [Background] Schievink WI, Maya MM, Pikul BK, Louy C. Spontaneous spinal cerebrospinal fluid leaks as the cause of subdural hematomas in elderly patients on anticoagulation. J Neurosurg. 2010 Feb;112(2):295-9. doi: 10.3171/2008.10.JNS08428. PMID 19199465
- [Background] Schievink WI, Moser FG, Maya MM. CSF-venous fistula in spontaneous intracranial hypotension. Neurology. 2014 Jul 29;83(5):472-3. doi: 10.1212/WNL.0000000000000639. Epub 2014 Jun 20. No abstract available. PMID 24951475
- [Background] Takahashi K, Mima T, Akiba Y. Chronic Subdural Hematoma Associated with Spontaneous Intracranial Hypotension: Therapeutic Strategies and Outcomes of 55 Cases. Neurol Med Chir (Tokyo). 2016;56(2):69-76. doi: 10.2176/nmc.oa.2015-0032. Epub 2015 Oct 21. PMID 26489406
- [Background] Yang W, Huang J. Chronic Subdural Hematoma: Epidemiology and Natural History. Neurosurg Clin N Am. 2017 Apr;28(2):205-210. doi: 10.1016/j.nec.2016.11.002. Epub 2017 Feb 1. PMID 28325454